CLINICAL TRIAL: NCT02684331
Title: Cardiac Magnetic Resonance Imaging in Type 2 Diabetes Mellitus: The Mechanisms of Cardiac Function and Perfusion Dysfunction
Brief Title: CMR in Type 2 Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: Slagelse Hospital (Other)
Responsible Party: Principal Investigator, Annemie Stege Bojer, Clinical assistant, Slagelse Hospital
Other Study IDs: SJ-490
Record Dates: First submitted 2016-02-08; First posted 2016-02-18 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2; Heart Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA-plasma Heparin-plasma Serum urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- T2DM
  Interventions: Other: Cardiac Magnetic Resonance Imaging (CMR); Other: Echocardiography; Other: Bood samples

INTERVENTIONS:
Other: Cardiac Magnetic Resonance Imaging (CMR) — An extensive explorative CMR protocol, including time/volume curves of LV and LA, rest and stress perfusion (with Adenosin) and time/volume curve of LA after chronotropic stress with Glycopyrrolate, further flow measurements and T1 mapping.
Other: Echocardiography — Standard measurements and strain.
Other: Bood samples — HbA1c, Glucose, Hgb, Creatinin, Sodium, Potassium, Total cholesterol, LDL cholesterol, HDL cholesterol, Free fatty acids, ALAT, Urinary albumin, NT-proBNP, ANP, suPAR, Copeptin, Proendothelin, proCNP, Soluble ST2, Galectin-3

SUMMARY:
The study will be performed as a cross-sectional survey. 300 Type 2 diabetes patients (T2DM), with or without known cardiovascular disease, will be recruited from the diabetes outpatient clinic, Slagelse Hospital. The patients will undergo echocardiography, Cardiac magnetic resonance imaging (CMR), clinical examination and will be asked to fill out questionnaires.

This study project sets out to answer the following hypotheses:

1. Patients with T2DM have an increased risk of developing diastolic dysfunction. Using CMR, the investigators wish to measure left ventricle peak filling rate and passive atrial emptying fraction as a measure of cardiac diastolic function. The investigators hypothesize that classic T2DM markers such as levels of urinary albumin excretion, retinopathy, autonomic neuropathy, hypertension, dyslipidemia, elevated HgbA1c, T2DM duration, etc. are associated with pathological findings by CMR.
2. Patients with T2DM have impaired left ventricle myocardial perfusion as determined by gadolinium contrast CMR. The investigators hypothesize that the classic markers and risk factors mentioned above, are associated with left ventricle myocardial hypoperfusion as determined by gadolinium contrast CMR.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient fully capable of informed consent
* Informed consent
* T2DM
* Age 18-80 (both years included)

Exclusion Criteria:

* Contraindications to CMR (pacemakers/ICD-units, cochlear implants)
* Lack of consent
* Atrial fibrillation
* eGFR < 30 ml/min/1,73m2 (only exclusion criteria for gadolinium contrast study)
* Women of childbearing potential who are not on acceptable contraception
* Severe claustrophobia (only contraindication for CMR but can undergo echocardiography and other examinations)
* Contraindications to adenosine: history of significant bronchial asthma, 2nd or 3rd degree AV-block, severe hypotension, long QT-syndrome, unstable angina pectoris, sinus node dysfunction, incompensated heart failure
* Contraindications to glycopyrrolate: closed-angle glaucoma, prostate hyperplasia, tachycardia, bladder atony, cardia insufficiency, non-congenital pylorus stenosis and gastroparesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 T2DM patients, with or without known cardiovascular disease, will be recruited from the diabetes outpatient clinic, Slagelse Hospital.
  The patients will be divided into groups depending on their diabetes complication status. Individual groups of patients with fx. +/- retinopathy, +/- autonomous neuropathy, +/- hypertension, normo-/mikro-/makroalbuminuria will be compared.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2016-01; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
On CMR; left ventricle peak filling rate (ml/s) | Cross-sectional so at baseline
  Measure for cardiac diastolic function; including measurements at rest and after glycopyrrolate chronotropic stress
On CMR, LV myocardial perfusion | Cross-sectional so at baseline
  Including measurements at rest and with Adenosin stress
On CMR; passive atrial emptying fraction (%) as a measure for cardiac diastolic function | Cross-sectional so at baseline
  Measure for cardiac diastolic function; including measurements at rest and after glycopyrrolate chronotropic stress

SECONDARY OUTCOMES:
Echocardiography | Cross-sectional so at baseline
  Systolic function
Blod samples | Cross-sectional so at baseline
  NT-proBNP, ANP, suPAR, Copeptin, Proendothelin, proCNP, Soluble ST2, Galectin-3
Echocardiography | Cross-sectional so at baseline
  Diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Soerensen, DM, Principal Investigator — Slagelse Hospital
Locations (1):
- The diabetes outpatient clinic, Slagelse Hospital, Denmark, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bojer AS, Sorensen MH, Madsen SH, Broadbent DA, Plein S, Gaede P, Madsen PL. The independent association of myocardial extracellular volume and myocardial blood flow with cardiac diastolic function in patients with type 2 diabetes: a prospective cross-sectional cohort study. Cardiovasc Diabetol. 2023 Mar 31;22(1):78. doi: 10.1186/s12933-023-01804-9. PMID 37004049
- [Derived] Bojer AS, Sorensen MH, Vejlstrup N, Goetze JP, Gaede P, Madsen PL. Distinct non-ischemic myocardial late gadolinium enhancement lesions in patients with type 2 diabetes. Cardiovasc Diabetol. 2020 Oct 22;19(1):184. doi: 10.1186/s12933-020-01160-y. PMID 33092588
- [Derived] Sorensen MH, Bojer AS, Jorgensen NR, Broadbent DA, Plein S, Madsen PL, Gaede P. Fibroblast growth factor-23 is associated with imaging markers of diabetic cardiomyopathy and anti-diabetic therapeutics. Cardiovasc Diabetol. 2020 Sep 30;19(1):158. doi: 10.1186/s12933-020-01135-z. PMID 32998751
- [Derived] Sorensen MH, Bojer AS, Pontoppidan JRN, Broadbent DA, Plein S, Madsen PL, Gaede P. Reduced Myocardial Perfusion Reserve in Type 2 Diabetes Is Caused by Increased Perfusion at Rest and Decreased Maximal Perfusion During Stress. Diabetes Care. 2020 Jun;43(6):1285-1292. doi: 10.2337/dc19-2172. Epub 2020 Mar 19. PMID 32193248
- [Derived] Sorensen MH, Bojer AS, Broadbent DA, Plein S, Madsen PL, Gaede P. Cardiac perfusion, structure, and function in type 2 diabetes mellitus with and without diabetic complications. Eur Heart J Cardiovasc Imaging. 2020 Aug 1;21(8):887-895. doi: 10.1093/ehjci/jez266. PMID 31642902